CLINICAL TRIAL: NCT02769910
Title: The Role of Pre-established Skin Inflammation on the Susceptibility to Histamine and Cowhage-induced Itch in Healthy Humans
Brief Title: Effects of High-concentration Topical Capsaicin on Histaminergic and Non-histaminergic Itch
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hjalte Holm Andersen (Other)
Responsible Party: Sponsor-Investigator, Hjalte Holm Andersen, MSc. Med., Phd. Stud., Aalborg University
Organization: Aalborg University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N-20160026
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cowhage (Other): Cowhage is used to induce non-histaminergic itch on the volar forearm at the locations treated with Capsaicin 24 Hours, Capsaicin 1 Hours and Qutenza Demo Patch.
  Interventions: Drug: Capsaicin 24 Hours; Drug: Capsaicin 1 Hour; Other: Qutenza Demo Patch
- Histamine (Other): Histamine is used to induce histaminergic itch on the volar forearm at the locations treated with Capsaicin 24 Hours, Capsaicin 1 Hour and Qutenza Demo Patch.
  Interventions: Drug: Capsaicin 24 Hours; Drug: Capsaicin 1 Hour; Other: Qutenza Demo Patch

INTERVENTIONS:
Drug: Capsaicin 24 Hours — Dermal patches for transdermal application of Capsaicin, applied for 24 hours
  Other Names: Qutenza
Drug: Capsaicin 1 Hour — Dermal patches for transdermal application of Capsaicin, applied for 1 hour
  Other Names: Qutenza
Other: Qutenza Demo Patch — Dermal patches mimicking active Qutenza patches. Used as control in comparison of Capsaicin efficacy. Applied for 24 hours.
  Other Names: Qutenza Demo

SUMMARY:
The purpose of this project is to investigate the effect of capsaicin-induced neurogenic inflammation with three different intensities on itch subsequently induced by histamine and cowhage. The hypothesis is that capsaicin-induced pre-established neurogenic inflammation significantly increases susceptibility to itch provocations with cowhage and histamine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Caucasian descent
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other drugs
* Previous or current neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* Current use of medications that may affect the trial
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Moles or tattoos in the area to be irradiated
* Exposure of the irradiated area to UV radiation (e.g., sun) 48 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Itch intensity | Assessed continuously at 0-10 minutes following itch provocation
  Rating of the perceived itch intensity on a visual analogue scale (VAS) App (Aalborg University) as displayed on a tablet computer with a sample rate of 1 Hz.

SECONDARY OUTCOMES:
Neurogenic inflammation | Assessed 11 minutes after itch provocation
  Neurogenic inflammation in the treated area is assessed using full-field laser perfusion imaging (FLPI)
Changes in sensitivity to touch-evoked itch | Assessed before, and at 12-15 minutes following itch provocation
  Three von Frey filaments are applied to the test area before and after itch provocation. Subjects report three NRS scores ('0-10', 'No itch-Worst imaginable itch') for itch induced by von Frey stimulation. Change is calculated by subtracting baseline mean from post-provocation mean NRS scores.
Wheal size | Assessed at 10 minutes following itch provocation
  Histamine wheal size is assessed by measuring the longest diameter of the wheal with a ruler, followed by measuring the orthogonal diameter. The mean of these diameters will represent the wheal size in diameter, reported in mm.
Pain intensity | Assessed continuously at 0-10 minutes following itch provocation
  Rating of the perceived pain intensity on a visual analogue scale (VAS) App (Aalborg University) as displayed on a tablet computer with a sample rate of 1 Hz.
Pain during capsaicin application | 24 hours after first application of capsaicin patch
  Peak and average numerical rating scale (NRS) scores ('0-10, 'no pain-worst imaginable pain') are reported by subjects for each patch.

CONTACTS AND LOCATIONS:
Locations (1):
- SMI, Aalborg, NJ, Denmark

IPD SHARING:
Plan to Share IPD: No